CLINICAL TRIAL: NCT06026696
Title: Cohorte de Maladies Neurovasculaires Prises en Charge à la Phase aiguë et Suivies à Lariboisière
Brief Title: Cohort of Neurovascular Diseases Treated in the Acute Phase and Followed at Lariboisière
Acronym: NERVAL
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221076
Record Dates: First submitted 2023-08-21; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-07

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for acute cerebrovascular pathology cerebrovascular disease
  Interventions: Other: follow-up

INTERVENTIONS:
Other: follow-up — Long term follow-up

SUMMARY:
Neurovascular diseases can cause ischaemic or haemorrhagic strokes. While the most common, such as atherosclerosis are widely studied, others are less well known, such as arterial dissections or cerebral angiopathies. What's more, most studies are limited to a few years' follow-up and the longer-term evolution of patients is less well assessed. Patient follow-up data available in routine practice and specific enrollment through the headache emergencies of the Lariboisière neurovascular intensive care unit (USINV) could provide a particularly rich resource.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥18 years
2. Patients admitted to the Neurovascular Intensive Care Unit with acute cerebrovascular disease OR Patients managed for acute cerebrovascular pathology with or without stroke by the Lariboisière neurology team.
3. No opposition from the patient to the research and for patients under guardianship or guardianship or lack of capacity to object (severe impairment of cognitive functions, dementia, etc.), no opposition from the legal representative.

Exclusion Criteria:

1. Patient refusing to take part in the study or refusal by the legal representative in the case of patients under guardianship or curatorship
2. Patient suffering from a rare neurovascular disease and being followed at the "Centre de référence des maladies vasculaires rares du cerveau et de l'oeil" (CERVCO)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated for acute cerebrovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2033-09 (Estimated); Study Completion 2038-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of a vascular event | Up to 5 years
  Vascular event is defined as : myocardial infarction, ischaemic or haemorrhagic stroke, recurrence of cerebrovascular disease, systemic embolism, congestive heart disease, vascular or non-vascular death during patient follow-up.

SECONDARY OUTCOMES:
Incidence of a vascular event | Up to 10 years
  Vascular event is defined as : myocardial infarction, ischaemic or haemorrhagic stroke, recurrence of cerebrovascular disease, systemic embolism, congestive heart disease, vascular or non-vascular death during patient follow-up.
Modified Rankin score | At 3 months
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 1 year
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 2 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 3 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 4 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 5 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 6 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 7 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 8 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 9 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Modified Rankin score | At 10 years
  The modified Rankin score is a 6 point disability scale varying between 0 to 5. The higher the score, the greater the disability.
Occurrence of intercurrent pathologies requiring specific treatment | Up to 10 years
  Pathologies are defined as : anxiety-depressive disorder, dementia, comititude, neoplasia, venous thromboembolism, haemorrhage, systemic disease, respiratory insufficiency
Obstetrical prognosis | Up to 10 years
  Incidence of pregnancies, complications, delivery methods
Incidence of death | Up to 10 years
  Age and causes of death
Prevalence of vascular risk factors | Up to 10 years
  Medical history, LDL (Low Density Lipoprotein), Tobacco, Arterial pressure, HbA1C (glycated hemoglobin)
Number of associated treatments | Up to 10 years
  Description of the types of treatment used
Number of adverse events | Up to 10 years
  Evaluation of treatment tolerance
Treatment adherence | Up to 10 years
Incidence of headaches | Up to 10 years

IPD SHARING:
Plan to Share IPD: Undecided